CLINICAL TRIAL: NCT00347789
Title: Efficacy of Transconjunctival Mitomycin-C in Needle Revisions of Failing Trabeculectomy
Brief Title: Effectiveness of a Procedure for Previously Failed Glaucoma Surgery
Status: Completed | Type: Observational
Sponsor: Glaucoma Research & Education Group (Other)
Collaborators: PharmaLogic Development, Inc. (Industry)
Other Study IDs: 11111
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Glaucoma
Keywords: glaucoma; trabeculectomy; filtering bleb revision; intraocular pressure; needling procedure; mitomycin C
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Glaucoma surgery- Bleb revision

SUMMARY:
Transconjunctival mitomycin-C in needle bleb revision may be an effective procedure to treat cases with a previously failed trabeculectomy. We will investigate approximately 100 consecutive cases with follow up of up to 9 years. We anticipate that this procedure is an effective, safe, and appropriate option for successful glaucoma treatment.

DETAILED DESCRIPTION:
The healing process after filtering surgery for glaucoma may cause an unsuccessful outcome for the trabeculectomy procedure. In order to control the rising intraocular pressure due to the failed trabeculectomy, medications may be restarted and/or filtering surgery may need to be repeated. Our primary research showed that transconjunctival mitomycin-C in needle bleb revision may be an effective procedure to control this situation.

This retrospective study will follow over 100 patients from May 1997 to May 2006. This long-term follow up will help assess the future role of this technique in glaucoma practices.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma
* Failed filtering procedures- defined as intraocular pressure exceeded target pressure thus inducing possible further optic nerve damage

Exclusion Criteria:

- Needling combined with other ocular surgical or laser treatments

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1997-05; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G. Iwach, MD, Principal Investigator — Glaucoma Reseach & Education Group
Locations (1):
- Glaucoma Center of San Francisco, San Francisco, California, United States